CLINICAL TRIAL: NCT00117507
Title: An Open Label, Safety and Tolerability Study of Deferasirox for Treatment of Transfusional Iron Overload in Low-Risk and INT-1 Myelodysplastic Patients
Brief Title: Study for the Treatment of Transfusional Iron Overload in Myelodysplastic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS02
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Myelodysplastic Syndromes; Iron Overload
Keywords: MDS; Myelodysplastic Syndrome; ICL-670; ICL-670 and Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Iron Overload | interventions — Deferasirox; Chelating Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): Participants received deferasirox 20mg/kg/day OD for 12 months. Deferasirox was taken every morning 30 minutes before breakfast, if possible consistently around the same time between 7:00 and 9:00 AM. The tablets was dropped into water or orange juice and gently stirred for 1 to 3 minutes until completely dispersed.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox
  Other Names: Chelator; Iron chelator

SUMMARY:
Thirty patients were to be enrolled and 24 patients were actually enrolled into this open-label, single-arm trial designed to assess the safety and tolerability of oral deferasirox in adult transfusion dependent myelodysplastic syndrome (MDS) patients with iron overload. Patients enrolled in this study had low or intermediate (INT-1) risk MDS per International Prognostic Scoring System (IPSS) criteria. All patients initiated treatment with 20mg/kg/day deferasirox.

Deferasirox were administered orally once per day for 12 months.

DETAILED DESCRIPTION:
Patients were screened for eligibility to determine if they meet all inclusion/exclusion criteria. The screening period were up to 4 weeks. Patient's baseline LIC will be determined non-invasively by means of MRI R2 analysis. In addition, blood and urine samples will be taken for the determination of baseline safety data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with low or intermediate (INT-1) risk MDS, determined via IPSS criteria, with transfusional iron overload. NOTE: Bone marrow morphology and cytogenetic studies completed within 3 months prior to screening can be used if the patient has been hematologically stable. Every attempt to obtain cytogenetics studies should be made; however, if there is culture failure, repeat marrow aspiration will not be mandated. In this case, RAEB with less than 11% marrow blasts will be accepted.
* Patients on chelation therapy at the time of screening required a 1-day wash out prior to the first dose of study drug.
* Age: greater than or equal to 18 years
* Serum ferritin:

  * For entry into the screening period: serum ferritin greater than or equal to 1000 µg/mL on at least two occasions, at least two weeks apart, during the prior year. Samples must be obtained in the absence of concomitant infection;
  * For enrollment into the study: serum ferritin greater than or equal to 1000 µg/mL at screening (via the central lab) obtained in the absence of concomitant infection
* A lifetime minimum of 20 previous packed red cell transfusions
* Life expectancy greater than or equal to 6 months
* Women must have a negative serum or urine pregnancy test and use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined by amenorrhea for at least 12 months).
* Able to provide written informed consent

Exclusion Criteria:

* Serum creatinine greater than 2 × upper limit of normal (ULN)
* ALT or AST greater than 5 × ULN.
* Clinical or laboratory evidence of active hepatitis B or hepatitis C (HBsAg in the absence of HBsAb -OR- HCV Ab positive with HCV RNA positive and ALT above the normal range)
* Significant proteinuria as indicated by a urinary protein/creatinine ratio greater than 0.5 mg/mg in a non-first void urine sample during screening (or alternatively in two of three samples obtained for screening)
* History of HIV positive test result (ELISA or Western blot)
* ECOG performance status greater than 2
* Uncontrolled systemic hypertension
* Unstable cardiac disease not controlled by standard medical therapy
* Third degree atrioventricular (AV) block or QT interval prolongation above the normal range
* History of clinically relevant ocular toxicity related to iron chelation
* Pregnancy or breast feeding
* Treatment with a systemic investigational drug within the past 4 weeks or a topical investigational drug within the past 7 days.
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following:

  * inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding;
  * major gastrointestinal tract surgery, such as gastrectomy, gastroenterostomy, or bowel resection;
  * pancreatic injury or pancreatitis or indications of impaired pancreatic function/injury, as indicated by abnormal lipase or amylase;
  * urinary obstruction or difficulty in voiding.
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Stanford University Medical Center, Stanford, California
  - Karmanos Cancer Center, Detroit, Michigan
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Greenberg PL, Koller CA, Cabantchik ZI, Warsi G, Glynos T, Paley C, Schiffer C. Prospective assessment of effects on iron-overload parameters of deferasirox therapy in patients with myelodysplastic syndromes. Leuk Res. 2010 Dec;34(12):1560-5. doi: 10.1016/j.leukres.2010.06.013. Epub 2010 Jul 8. PMID 20615548
- See also: Results for CICL670AUS02 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants at 3 centers in United States.
Pre-assignment Details: A total 24 participants were enrolled in the study of which 9 participants completed the study and 15 participants discontinued from the study.
Groups:
- Deferasirox: Participants received deferasirox 20mg/kg/day OD (Once Daily) per day for 12 months. Deferasirox was taken every morning 30 minutes before breakfast, if possible consistently around the same time between 7:00 and 9:00 AM. The tablets was dropped into water or orange juice and gently stirred for 1 to 3 minutes until completely dispersed.
Period: Overall Study
Arm/Group | Deferasirox
Started | 24
Completed | 9
Not Completed | 15
Not completed — Adverse Event | 4
Not completed — Abnormal laboratory values | 3
Not completed — Unsatisfactory therapeutic effect | 1
Not completed — Patient withdrew consent | 4
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all patients who were registered in the study, whether or not they received treatment.
Groups:
- Deferasirox: Participants received deferasirox 20mg/kg/day OD per day for 12 months.
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study. Any sign or symptom that occured from first dose of study treatment until end of study treatment.
Time Frame: Up To Week 52
Population: The safety set consisted of all participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
Participants
  Adverse events | 24
  Serious adverse events | 11

2. Secondary Outcome: Absolute Change in Serum Ferritin From Baseline to Week 52
Description: Absolute change in serum ferritin after start of treatment with Deferasirox (ICL670).
Time Frame: Baseline to Week 52
Population: Intent-to-treat (ITT) population consisted of all participants who were registered in the study, whether or not they received treatment.
Measure: Mean (Standard Deviation); unit: μg/L (microgram/litre)
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
μg/L (microgram/litre)
  Baseline | 3847.6 (2854.54)
  Week 52/EOS (end of study): number analyzed (Participants) | 19
  Week 52/EOS (end of study) | -729.8 (2749.35)

3. Secondary Outcome: Absolute Change in Liver Iron Concentration (LIC) From Baseline to End of Study
Description: LIC was assessed using magnetic resonance imaging (MRI) mean liver proton transverse relaxation rates (R2).
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg iron (Fe) per gram of dry weight (dw)
Groups:
- Deferasirox: Participants received deferasirox 20mg/kg/day OD per day for 12 months. Deferasirox was taken every morning 30 minutes before breakfast, if possible consistently around the same time between 7:00 and 9:00 AM. The tablets was dropped into water or orange juice and gently stirred for 1 to 3 minutes until completely dispersed.
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
mg iron (Fe) per gram of dry weight (dw)
  Baseline | 20.64 (9.747)
  Week 52/EOS: number analyzed (Participants) | 13
  Week 52/EOS | -4.50 (12.995)

4. Secondary Outcome: To Evaluate Change in Transfusion Requirements
Description: Change in transfusion requirements from baseline.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: blood tranfusions
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
blood tranfusions
  Number of Transfusions per Patient | 15.5 (9.46)
  Number of Units of Blood Transfused per Patient | 34.0 (24.65)

5. Secondary Outcome: Absolute Change in Serum Erythropoietin
Description: Absolute Change in Serum Erythropoietin from baseline.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU (international unit)/L (litre)
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
IU (international unit)/L (litre)
  Baseline | 646.50 [46.9 to 3779.0]
  Week 52/EOS: number analyzed (Participants) | 19
  Week 52/EOS | -79.00 [-949.0 to 1091.0]

6. Secondary Outcome: Absolute Change in Urinary Hepcidin
Description: Absolute Change in Urinary Hepcidin from baseline
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng (nanogram)/mg (milligram) creatinine
Arm/Group | Deferasirox
Number analyzed (Participants) | 17
ng (nanogram)/mg (milligram) creatinine
  Baseline | 327.63 [17.5 to 1993.1]
  Week 52/EOS: number analyzed (Participants) | 9
  Week 52/EOS | 67.32 [-819.4 to 1100.1]

7. Secondary Outcome: Absolute Change in Transferrin Saturation
Description: Transferrin Saturation was assessed using magnetic resonance imaging (MRI) mean liver proton transverse relaxation rates (R2)
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of transferrin saturation
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
percentage of transferrin saturation
  Baseline | 59.3 (7.24)
  Week 52/EOS (Change from baseline): number analyzed (Participants) | 19
  Week 52/EOS (Change from baseline) | 8.6 (21.19)

8. Secondary Outcome: Labile Plasma Iron (LPI)
Description: LPI represents the component of non-transferrin bound iron and is an indicator of iron overload. The outcome was reported as LPI Unit, where, 1 LPI unit = the quantity of reactive oxygen species produced by approximately 1.5 μM Fe.
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: LPI Unit
Arm/Group | Deferasirox
Number analyzed (Participants) | 24
LPI Unit
  Baseline | 0.70 (0.638)
  Week 52/EOS | 0.22 (0.460)

ADVERSE EVENTS:
Time Frame: Adverse events were collected From Start of the Study up to EOS (Week 52). The safety set consisted of all participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.
Arm/Group | Deferasirox
All-Cause Mortality (participants affected / at risk) | 3/24
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=24)
Splenic infarction (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Left ventricular hypertrophy (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 2
Chills (General disorders) | 1
Concomitant disease progression (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 4
Cholecystitis acute (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=24)
Leukocytosis (Blood and lymphatic system disorders) | 1
Monocytosis (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dilatation atrial (Cardiac disorders) | 1
Dilatation ventricular (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctival discolouration (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 15
Flatulence (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Odynophagia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Concomitant disease progression (General disorders) | 1
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 1
Malaise (General disorders) | 1
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Hepatomegaly (Hepatobiliary disorders) | 3
Jaundice (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 3
Catheter related infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Excoriation (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate irregular (Investigations) | 1
Lipase increased (Investigations) | 1
Weight decreased (Investigations) | 6
Weight increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No